CLINICAL TRIAL: NCT04433338
Title: The PREBA Study: Effect of Preoperative Weight Loss With a 14-day Low-calorie Diet on Surgical Procedure and Outcomes in Patients Undergoing RYGB Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL70092.081.19
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery; Morbid Obesity
Keywords: Bariatric surgery; Morbid Obesity; Weight Loss; Diet; RYGB
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will follow a low-calorie diet during 14 days before undergoing surgery. The diet will consist of both meal replacements and regular foods.
  For women, the diet provides ± 900 kcal, 50 grams of carbohydrates, 85 grams of protein, 30 grams of fat and 25 grams of fibres.
  For men, the diet provides ± 1000 kcal, 55 grams of carbohydrates, 100 grams of protein, 30 grams of fat and 30 grams of fibres.
  Interventions: Other: 14-day Low Calorie Diet
- Control group (No Intervention): Participants in the control group can eat according to the standard nutritional advices provided by their dietitian. These advices are intended to educate participants on the recommended eating pattern after surgery.

INTERVENTIONS:
Other: 14-day Low Calorie Diet — Participants will be asked to:
  * Use 4 (women) or 5 (men) Modifast meal replacements per day.
  * Daily consume a minimum of 250 grams of (raw) vegetables without dressing.
  * Daily consume 100 grams of lean meat/fish/meat analogues.
  * Daily consume two spoons of liquid oil
  * Daily drink at least 2.0 litres of water, coffee or tea without added sugar or milk, bouillon or sugar-free drinks.
  Arms: Intervention group

SUMMARY:
Bariatric guidelines recommend preoperative weight loss of 5% to reduce the risk of surgical complications. However, results in the literature on the improvement of surgical procedure and outcomes are still conflicting.

This study aims to evaluate the effect of preoperative weight loss by means of a 14-day low-calorie diet in bariatric patients on operative time, the ease of the Roux-en-Y gastric bypass (RYGB) procedure and long-term weight loss in a real-life experimental setting.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary RYGB surgery (meeting all criteria + approval of surgeon)
* Able to prepare the meal replacements at home

Exclusion Criteria:

* Undergoing another bariatric procedure than primary RYGB.
* Diabetes Mellitus
* Contraindication for the usage of Modifast meal replacements:

  * Allergy or intolerance to any substance in the used meal replacements (Soy, milk, gluten, egg, peanuts, nuts and seeds)
  * Veganism
  * Kidney failure (GFR < 90 ml/min/1.73m2), liver failure or cardiac insufficiency
  * A heart attack (myocardial infarct) in the past twelve months
  * Cancer
  * Hypokalaemia: serum potassium level <3.4 mmol/l
  * Phenylketonuria & Porphyria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Operative time of the RYGB procedure | surgery
  Duration of the surgical procedure, retrieved from the electronic medical record

SECONDARY OUTCOMES:
Ease of the RYGB procedure | surgery
  Ten aspects of the RYGB procedure will be scored on a 5-point Likert scale. The total score can range from 10 to 50, with 10 being the easiest.
  The ten aspects include:
  * Exerting force on instruments (1=very low, 5= very high)
  * Difficulty of moving the liver (1=very easy, 5=very difficult)
  * Size of the liver (1=very small, 5= very large)
  * Size of omentum (1=very small, 5= very large)
  * Difficulty of approaching pouch (1=very easy, 5=very difficult)
  * Accessibility of Treitz ligament (1=very easy, 5=very difficult)
  * Difficulty of creating pouch (1=very easy, 5=very difficult)
  * Difficulty of measuring small intestine (1=very easy, 5=very difficult)
  * Difficulty of entero-entero connection (1=very easy, 5=very difficult)
  * Difficulty of abdominal wall hernia repair (1=very easy, 5=very difficult)
Appearance of the patient's liver | surgery
  Includes four images of the liver in different stages (1= healthy, 2= fatty liver, 3= fatty liver with inflammation, 4= liver cirrhosis). Surgeons will be asked to choose the image that best matches the appearance of the patient's liver.
Post-operative weight loss | 4 weeks, 3, 6 months and 1, 2, 3, 4, 5 years after surgery
  Body weight measurements to assess weight loss after surgery

OTHER OUTCOMES:
Feasibility of the diet | During the 14-day intervention period
  Feasibility will be assessed via questionnaires
Compliance of the diet | During the 14-day intervention period
  Compliance will be assessed via food records
Complication rate | First 30 days post-surgery
  All short term complications during the first 30 days will be recorded and classified according to the Clavien-Dindo classification
Wound healing | 4 weeks
  Degree of wound healing post-surgery will be checked based on appearance on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Hazebroek, MD, PhD, Principal Investigator — Vitalys, part of Rijnstate hospital/Wageningen University
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No